CLINICAL TRIAL: NCT05326906
Title: The Prediction Biomarkers of Survival Outcome for Severe Immune-related Hepatitis in Lung Cancer
Brief Title: The Prediction Biomarkers of Survival Outcome for Severe Immune-related Hepatitis
Status: Completed | Type: Observational
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Director, Head of Medical Oncology, Principal Investigator, Clinical Professor, Hunan Province Tumor Hospital
Other Study IDs: STEM
Record Dates: First submitted 2022-03-24; First posted 2022-04-14 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — tissue sample and blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: PD-1/PD-L1 inhibitors — PD-1/PD-L1 inhibitors (the dosage calculation according to dosing instructions)

SUMMARY:
Immune checkpoint inhibitors have revolutionized lung cancer (LC) treatment, demonstrating a significant improvement in overall survival. However high-grade immune-related adverse events (irAEs) may result in harmful and serious clinical outcomes, even death. Immune-related hepatitis (IRH) is a potentially serious complication of checkpoint blockade, with an incidence of 5%-10% for ICIs monotherapy, including 1%-2% with grade 3 or higher. Therefore, it is particularly important to explore new and better prognostic and predictive biomarkers for IRH.

ELIGIBILITY:
Inclusion Criteria:

* The lung cancers were diagnosed by pathological evaluation.
* The PD-1/PD-L1 inhibitors were administered in all patients.
* Grade 3-5 immune-related hepatitis had occurred.
* The pre-treatment tissues or peripheral blood were available.

Exclusion Criteria:

* The pathological type was not lung cancers.
* Grade 1-2 immune-related hepatitis would be excluded.
* The any-grade hepatitis were induced by chemotherapy or virus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with immuntherapy underwent severe Immune-related Hepatitis
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Immune-Related Hepatitis | 2 years
  Number of participants with Grade 3-4 IRH graded by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Number of Participants Deaths | 2 years
  Number of participants with Grade 3-4 immune-related hepatitis by CTCAE 4.0 who still died after the corticosteroid (2mg/kg) and/or mycophenolate mofetil treatment.

SECONDARY OUTCOMES:
Number of Participants with Laboratory Abnormalities in Liver Tests | 2 years
  Number of participants with laboratory liver tests based on Hunan Cancer hospital to determine the safety of immunotherapy. The number of participants with the following laboratory abnormalities from on-treatment evaluations will be summarized: ALT or AST >5-20 ULN, and > 20 x ULN;Total bilirubin > 3-10 ULN and > 10 x ULN

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Cancer hospital, Changsha, Hunan, China